CLINICAL TRIAL: NCT06320795
Title: Studio Prospettico Per la Validazione Clinica Del Dispositivo Medico Indossabile Soundi
Brief Title: Prospective Study for the Clinical Validation of the Soundi Wearable Medical Device
Acronym: SOUNDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biocubica srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IT-MF-000031905
Record Dates: First submitted 2024-03-07; First posted 2024-03-20 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-03

CONDITIONS: OSA

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soundi (Experimental): Soundi device compared to overnight polysomnography
  Interventions: Device: SOUNDI

INTERVENTIONS:
Device: SOUNDI — Continuous monitoring of vital signs for diagnosis and follow-up of sleep-disordered breathing in adults.

SUMMARY:
This is a pre-marketing, single-centre, prospective clinical trial with the aim of comparison the effectiveness and safety of the SOUNDI medical device compared to polysomnography in detecting parameters for the diagnosis of obstructive sleep apnea (OSA) syndrome in subjects with suspected diagnosis of sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to understand the nature of the study and to give free informed consent
* Must be over 20 and referred by medical staff for an overnight assessment for suspected sleep apnea

Exclusion Criteria:

* Pregnancy
* Pacemaker wearer
* Allergies to any material of the device

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of the clinical diagnosis of OSA | 6 Months
  To evaluate the accuracy of the clinical diagnosis of OSA assisted by the home sleep study with SOUNDI against the clinical diagnosis assisted by the PSG as the reference standard.
To evaluate the agreement between the Apnea Hypopnea Index (AHI) from the home sleep study with SOUNDI and the home sleep study with polysomnography (PSG) | 6 Months
  To evaluate the agreement between the AHI from the home sleep study with SOUNDI and the home sleep study with PSG in patients being referred to sleep clinics with suggestive OSA symptoms.

SECONDARY OUTCOMES:
Patient satisfaction | Day 1
  Patient satisfaction were determined by interview.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Lombardi, Prof., Principal Investigator — Istituo Auxologico Italiano
Locations (1):
- Ambulatorio del Sonno- Istituto Auxologico Italiano IRCCS - Ospedale San Luca, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT06320795/Prot_000.pdf